CLINICAL TRIAL: NCT03495713
Title: RadVax for Relapsed/Refractory Hodgkin's Lymphoma: A Phase II Trial of Nivolumab + Low Dose Radiotherapy for Incomplete Responders
Brief Title: Lymphoma RadVax LYMPHOMA: A PHASE II TRIAL OF NIVOLUMAB + LOW DOSE RADIOTHERAPY FOR INCOMPLETE RESPONDERS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04418
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Subjects will receive initial treatment with the immunomodulatory agent, nivolumab, followed by low-dose (4 Gy x 2) involved-site radiotherapy in subjects with less than an anatomic CR after the first restaging scan. Patients with anatomic CR will continue nivolumab alone without radiotherapy. Eligible patients will have r/r disease with at least 2 sites of measurable disease, and must be eligible for treatment with nivolumab.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3 mg/kg will be administered on day 1 (pre-response assessment week 0) and on day 1 and continued per standard of care and institutional practices. A
  Other Names: Opdivo

SUMMARY:
This is a Phase II single-arm, single-site, open label clinical trial with r/r HL patients, aimed to determine whether a RadVax approach using low-dose RT added to nivolumab can improve response among patients who do not achieve a CR to nivolumab alone. The long-term goal is to develop an effective regimen for r/r HL patients.

DETAILED DESCRIPTION:
Nivolumab 3 mg/kg will be administered on day 1 (pre-response assessment week 0) and on day 1 and continued per standard of care and institutional practices. At the week 1 biomarker collection, research FDG PET/CT will be performed to assess for FDG "flare." At week 8-12, PET/CT will be performed for the first response assessment. If a complete anatomic response is seen, nivolumab monotherapy will be continued on day 1 and continued per standard of care and institutional practices.

By contrast, if at week 8 less than a complete anatomic response is seen, radiotherapy to 4 Gy x 2 fractions will be administered (post-response assessment week 0). The patient will be evaluated by a radiation oncologist while on treatment, and toxicities will be recorded. Nivolumab will be continued on day 1 and continued per standard of care and institutional practices.

In either scenario, a second response assessment will be conducted ~8-12 weeks after the first response assessment. In either scenario, nivolumab monotherapy will be continued at the discretion of the treating medical oncologist.

If there is less than CR post-RT and there is an additional untreated non-target lesion that can be followed, radiotherapy can again be administered when disease progresses to a previously untreated lesion, after which the patient will continue on the post-RT follow-up algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Hodgkin lymphoma for whom nivolumab is clinically indicated.
* Relapsed/refractory disease.
* ≥2 sites of measurable disease, at least one outside of intended RT fields.
* Age ≥ 18 years.
* ECOG performance status of 0-2.
* Standard laboratory criteria for hematologic, and biochemical, and urinary indices within a range that, in the opinion of the physician, clinically supports enrollment of the subject on the trial.
* Patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial.
* Ability to provide written informed consent.

Exclusion Criteria:

* Subjects with contraindications to immune checkpoint therapy, as follows:
* Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity.
* Prior organ allograft or allogeneic bone marrow transplantation.
* Subjects with contraindications to immune checkpoint therapy, as follows:
* Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity.
* Prior organ allograft or allogeneic bone marrow transplantation.
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Active autoimmune disease, except for vitiligo, type 1 diabetes mellitus, asthma, atopic dermatitis, or endocrinopathies manageable by hormone replacement; other autoimmune conditions may be allowable at the discretion of the principal investigator.
* Condition requiring systemic treatment with either corticosteroids.
* Systemic steroids at physiologic doses (equivalent to dose of oral prednisone 10 mg) are permitted. Steroids as anti-emetics for chemotherapy are strongly discouraged
* Intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted.
* Pregnant women, women planning to become pregnant and women that are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Plastaras, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 29 [20 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Overall complete response rate as determined by re-staging scan
Time Frame: 25 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 7
Participants | 7
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; Descriptive analysis only based limited enrollments

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=7)
Non-cardiac chest pain (Cardiac disorders) | 1 (1)
Pregnancy loss (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anaphylaxis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT03495713/Prot_SAP_000.pdf